CLINICAL TRIAL: NCT05506605
Title: Open-label, Single-arm, Unicenter and Pilot Study of a Switch Strategy From Etravirine (ETR) to Doravirine (DOR) in Virologically-Suppressed HIV-1 Infected Adults With ETR-Resistance
Brief Title: Switch Strategy From Etravirine (ETR) to Doravirine (DOR) in Virologically-Suppressed HIV-1 Infected Adults With ETR-Resistance
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Principal Investigator, Anna Cruceta, Medical Coordinator, Fundacion Clinic per a la Recerca Biomédica
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DoRSwitch.21
Record Dates: First submitted 2022-07-22; First posted 2022-08-18 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: HIV-1-infection
Keywords: HIV; Doravirine; Etravirine
MeSH Terms: interventions — doravirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Switch from Etravirine to Doravirine (Experimental): Switch from etravirine to Doravirine (Pifeltro) 100 mg each day
  Interventions: Drug: Doravirine 100Mg Tab

INTERVENTIONS:
Drug: Doravirine 100Mg Tab — Switch from Etravirine to Doravirine

SUMMARY:
Phase IV, open-label, single arm, unicenter and pilot study on virologically suppressed HIV infected adults with ETR resistance, to assess the efficacy of a Switch strategy from Etravirine (ETR) to Doravirine (DOR).

ELIGIBILITY:
Inclusion Criteria:

* HIV-1-infected subjects with age ≥18 years old.
* Desire of the patient to simplify their ART-regimen.
* Having plasma HIV-1 RNA < 50 copies/mL during at least the previous 24 weeks.
* Currently receiving an ETR-containing regimen (unchanged during the previous 24 weeks).
* Documented pooled/historical genotype or GRT in pro-viral DNA must show the presence of 103N and/or 181C and/or 190A and/or 100I and/or 138K/A.

Exclusion Criteria:

* Documented pooled/historical genotype or GRT in pro-viral DNA of any DOR-DRM (Mutations V106A, Y188L, and M230L, and combinations of V106A and L234I; V106A and F227L and L234I; and V106A and 190A and F227L).
* Pregnant, breastfeeding women, women with a positive pregnancy test at the time of screening, sexually active fertile women wishing to conceive or unwilling to commit to contraceptive methods, for the duration of the study and until 4 weeks after the last dose of study medication. All women are considered fertile unless they have undergone a sterilizing surgery or are over the age of 50 with spontaneous amenorrhea for over 12 months prior to study entry.
* Active tuberculosis infection.
* Any clinical condition or therapy that, in the opinion of the Investigator, would make the individual unsuitable for the study or unable to comply with the dosing requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with confirmed HIV viral load>50 copies/mL | at week 24
  Measured by blood HIV viral load

SECONDARY OUTCOMES:
Percentage of participants with HIV viral load>50 copies/mL | at week 12 and 48
  Measured by blood HIV viral load
Percentage of participants with HIV viral load<50 copies/mL | at week 12, 24 and 48
  Measured by blood HIV viral load
Changes in CD4, CD8 cell counts and ratio CD4/CD8 | at 48 weeks
  Measured by blood CD4, CD8 and CD/4/CD8 ratio
Incidence of Treatment-Emergent adverse events and serious adverse events | at week 48
  Measured by numer of AEs and SAEs related to the treatment
AUC during the dose interval (AUC0-24) of DRV/r and DRV/c with DOR | at weeks 2 and 4
Maximum concentrations (Cmax) of DRV/r and DRV/c with DOR | at weeks 2 and 4
Concentrations at the end of the dosing interval (C24) of DRV/r and DRV/c with DOR | at weeks 2 and 4
Elimination half-life (t1/2) of DRV/r and DRV/c with DOR | at weeks 2 and 4

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic i Provincial de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No